CLINICAL TRIAL: NCT02458716
Title: Feasibility of Cytoreductive Prostatectomy in Men Newly Diagnosed With Metastatic Prostate Cancer
Brief Title: Cytoreductive Prostatectomy in Treating Patients With Newly Diagnosed, Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Isaac Yi Kim, MD, PhD, MBA, Associate Professor, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro20140001022; NCI-2015-00384 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20140001022 (Other: IRB Number); 081403 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2015-04-06; First posted 2015-06-01 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Prostate Carcinoma; Metastatic Prostatic Adenocarcinoma; Prostate Carcinoma Metastatic to the Bone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery followed by hormone therapy (ADT) (Experimental): Patients undergo Robotic Assisted Radical Prostatectomy (RARP) or conventional open retropubic radical prostectomy (RRP). Immediately following surgery, patients receive the standard systemic androgen deprivation therapy.
  Interventions: Procedure: Robotic Assisted Radical Prostatectomy; Procedure: Conventional open retropubic radical prostectomy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: ADT (androgen deprivation therapy) (i.e. leuprolide) plus an androgen receptor inhibitor (i.e. bicalutamide)

INTERVENTIONS:
Procedure: Robotic Assisted Radical Prostatectomy — Undergo RARP
Procedure: Conventional open retropubic radical prostectomy — Undergo conventional open RRP
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: ADT (androgen deprivation therapy) (i.e. leuprolide) plus an androgen receptor inhibitor (i.e. bicalutamide) — LHRH agonist or antagonist (i.e. leuprolide) plus an androgen receptor inhibitor (i.e. bicalutamide)
  Other Names: Hormone therapy

SUMMARY:
This phase I trial studies the side effects of cytoreductive prostatectomy in treating patients with newly diagnosed prostate cancer that has spread from the primary site to other places in the body. Cytoreductive prostatectomy is a type of surgery that removes the prostate and as much of the tumor as possible. When combined with hormone therapy, robotic assisted radical prostatectomy (RARP) or conventional open retropubic radical prostatectomy (RRP) may prolong survival in patients with prostate cancer that has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of cytoreductive prostatectomy (to remove as much of the primary cancer as possible) in men with newly diagnosed clinical T1-3N1M0 or T1-3N0M1a-b prostate cancer (herein, collectively referred to as metastatic prostate cancer).

SECONDARY OBJECTIVES:

I. Time to prostate specific antigen (PSA) nadir and castration resistance following cytoreductive prostatectomy and subsequent standard systemic therapy, androgen deprivation.

OUTLINE:

Patients undergo RARP or conventional open RRP. Immediately following surgery, patients receive standard systemic androgen deprivation therapy.

After completion of study treatment, patients are followed up every 90 days for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate
* Evidence of lymph node or bone metastasis by magnetic resonance imaging (MRI)/computed tomography (CT), bone scan, or biopsy (N1Mx or NxM1)
* Give informed consent
* Clinical stage T3 or less (pelvic MRI shows no rectal and ureteral invasion)
* Cleared by the primary medical doctor for surgery
* No prior systemic therapy for metastatic prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Refuses to give informed consent
* Refuses or is unable to have pelvic MRI
* Clinical stage T4 (pelvic MRI shows rectal and/or ureteral invasion)
* Deemed a poor surgical risk per primary medical doctor
* Received prior therapeutic intervention for metastatic prostate cancer
* Known spinal cord compression or brain or liver metastasis
* Deep vein thrombosis (DVT)/pulmonary embolism (PE) in the past 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Rate of major peri-operative complications defined as Clavien-Dindo grade III or higher | Within 90 days after cytoreductive prostatectomy
  Rate will be calculated for the primary end point, and one-sided Binomial test will be used to compare the rate to the hypothesized value. Descriptive statistics will be provided. Any further statistical analysis deemed necessary to calculate significant findings will be done with the assistance of the Rutgers Cancer Institute of New Jersey Biostatistics Section.

SECONDARY OUTCOMES:
Time to PSA nadir | Up to 3 years
  Time to event data will be analyzed using the Kaplan-Meier product limit method. Descriptive statistics will be provided. Any further statistical analysis deemed necessary to calculate significant findings will be done with the assistance of the Rutgers Cancer Institute of New Jersey Biostatistics Section.
Time to rising PSA while on the standard androgen deprivation therapy | Up to 3 years
  Time to event data will be analyzed using the Kaplan-Meier product limit method. Descriptive statistics will be provided. Any further statistical analysis deemed necessary to calculate significant findings will be done with the assistance of the Rutgers Cancer Institute of New Jersey Biostatistics Section.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Kim, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - City of Hope National Medical Center (COH), Duarte, California
  - University of California, Irvine (UCI), Orange, California
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey